CLINICAL TRIAL: NCT00003148
Title: Phase II Study of the Efficacy of rH Interleukin-2 in Patients With Slowly Progressing Acute Myelogenous Leukemia (AML) and With Limited Bone Marrow Blastosis After Autologous Stem Cell Transplantation or Chemotherapy
Brief Title: Interleukin-2 in Treating Patients With Relapsed or Refractory Acute Myelogenous Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-06964; EORTC-06964
Record Dates: First submitted 1999-11-01; First posted 2004-04-23 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Leukemia
Keywords: recurrent adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin

SUMMARY:
RATIONALE: Interleukin-2 may stimulate a person's white blood cells to kill acute myelogenous leukemia cells.

PURPOSE: Phase II trial to study the effectiveness of interleukin-2 in treating patients with acute myelogenous leukemia that has relapsed following previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the therapeutic activity of interleukin-2 (IL-2) in patients with slowly progressing acute myeloid leukemia with limited bone marrow blastosis either in first relapse after autologous bone marrow or peripheral blood stem cell transplantation, or with more advanced disease (i.e., refractory to chemotherapy regimens). II. Characterize the acute side effects of IL-2 in these patients.

OUTLINE: This is an open label, nonrandomized, multicenter study. Patients are stratified into two categories of prior failed treatments (first relapse after autologous bone marrow or peripheral blood stem cell transplantation vs first or subsequent relapse either refractory to or not eligible for further conventional treatment). Interleukin-2 (IL-2) is administered as a continuous intravenous infusion on 5 consecutive days at daily escalating doses for the first cycle. When the individual maximum tolerated dose (MTD) has been determined, 3 more cycles are given at the MTD. There are 3 days of rest between each treatment cycle. After the induction phase, maintenance cycles of IL-2 are administered starting 4 weeks after the last induction treatment. Maintenance cycles of IL-2 are administered subcutaneously on 5 consecutive days every 4 weeks for 2 years, and subsequently every other month for a maximum of 3 years. Treatment continues until disease progression or unacceptable toxicity for a maximum of 5 years. Patients are followed every 4 weeks during the first 2 years, then every 8 weeks during the next 3 years or until documented progression, and then every 3 months until death.

PROJECTED ACCRUAL: A maximum of 86 (57 transplanted; 29 patients nontransplanted) patients will be accrued into this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed acute myeloid leukemia (AML) that has relapsed after prior treatment(s) Slowly progressing disease as defined by bone marrow blasts of greater than 5% and less than 30% confirmed by at least 2 marrow aspirates taken 2 weeks apart Must be in either: First relapse after autologous bone marrow or peripheral blood stem cell transplantation OR First or subsequent relapse either refractory to or not eligible for further conventional treatment regimens

PATIENT CHARACTERISTICS: Age: 18 to 60 Performance status: WHO 0-2 Life expectancy: At least 3 months Hematopoietic: Not specified Hepatic: Bilirubin less than 2 times normal Renal: Creatinine less than 2 times normal Cardiovascular: Ejection fraction normal Pulmonary: PLCO diffusion greater than 60% Other: No active uncontrolled infections No other progressive malignant disease Not a poor medical risk because of nonmalignant systemic disease

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics Endocrine therapy: No concurrent steroids Radiotherapy: Not specified Surgery: Not specified Other: No concurrent indomethacin No other concurrent anticancer or investigational therapy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 86 (Estimated)
Dates: Start 1997-10; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roel Willemze, MD, PhD, Study Chair — Leiden University Medical Center
Locations (10):
- Innsbruck Universitaetsklinik, Innsbruck, Austria
- Belgium (2):
  - Institut Jules Bordet, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
- University Hospital Rebro, Zagreb, Croatia
- France (2):
  - Hotel Dieu de Paris, Paris
  - Institut Gustave Roussy, Villejuif
- Italy (2):
  - Ospedale San Eugenio, Rome
  - Azienda Policlinico Umberto Primo, Rome
- Netherlands (2):
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen